CLINICAL TRIAL: NCT01362140
Title: A Multicenter, Randomised, Double-blind, Placebo-controlled Study of Darbepoetin Alfa for the Treatment of Anaemic Subjects With Low or Intermediate-1 Risk Myelodysplastic Syndrome (MDS)
Brief Title: Darbepoetin Alfa in Patients With Anemic Low or Intermediate-1 Risk Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 20090160; 2009-016522-14 (EudraCT Number)
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: MDS
Keywords: Randomized; Darbepoetin alfa; Myelodysplastic Syndromes; Placebo-controlled; low risk MDS; intermediate-1 risk MDS; International Prognostic Scoring System
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Darbepoetin alfa (Experimental): Participants received darbepoetin alfa 500 µg every three weeks (Q3W) for 24 weeks in the double-blind treatment period, and continued to receive darbepoetin alfa 500 µg Q3W during the active treatment period for an additional 48 weeks.
  Interventions: Drug: Darbepoetin alfa
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injection every 3 weeks (Q3W) for 24 weeks during the double-blind treatment period. From week 25 participants received darbepoetin alfa 500 µg Q3W during the active treatment period for 48 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Darbepoetin alfa — Administered by subcutaneous injection every 3 weeks
  Other Names: Aranesp
  Arms: Darbepoetin alfa
Drug: Placebo — Administered by subcutaneous injection every 3 weeks
  Arms: Placebo

SUMMARY:
The primary objective was to assess the superiority of darbepoetin alfa versus placebo on the incidence of red blood cell transfusions during the 24-week double-blind treatment period in anemic patients with low or intermediate-1 risk MDS.

DETAILED DESCRIPTION:
This study consists of a 3-week screening period, a 24-week double-blind treatment period, and a 48-week active treatment period and the long-term follow-up period.

An end of treatment period (EOTP) visit occurs at week 25, or 3 weeks after last dose of investigational product (IP) for participants who withdraw from the study. After entering the active treatment period, an end of active treatment period (EOATP) visit occurs at week 72 / 73, or 3 weeks after the last dose of darbepoetin alfa.

Long-term follow-up (LTFU) will occur every 26 weeks (± 4 weeks) from the EOATP visit (or EOTP visit if the participant does not enter the active treatment period) and will continue for a minimum of 3 years from the first dose of IP. Follow-up may occur through clinic visit or telephone contacts. Information on the participant's survival and progression to AML status will be collected during LTFU.

ELIGIBILITY:
Inclusion Criteria:

* Low or intermediate-1 risk MDS patients per International Prognostic Scoring System (IPSS) at the time of randomisation, as determined by complete blood count (CBC) during screening and bone marrow examination and marrow cytogenetic analysis performed within 16 weeks prior to randomisation. Subject cannot have been rendered low or intermediate-1 risk by prior disease modifying therapy. Bone marrow slides must be available for centralized review at any time throughout the study
* World Health Organization (WHO) classification of refractory anemia (RA), refractory anemia with ring sideroblasts (RARS), refractory cytopenias with multilineage dysplasia (RCMD), MDS-unclassified (MDSU), MDS with isolated del(5q) (5q- syndrome) or refractory anaemia with excess blasts-1 (RAEB-1)
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 assessed during screening
* Haemoglobin level ≤ 10.0 g/dL as assessed by the local laboratory; sample obtained within 7 days prior to randomisation (retest during screening is acceptable)
* Adequate transferrin saturation (Tsat) (≥ 15%) and serum ferritin (≥ 10 ng/mL) as assessed by the central laboratory during screening (supplementation and retest during screening is acceptable)
* Adequate serum folate (≥ 4.5 nmol/L [≥ 2.0 ng/mL]) or RBC folate (≥ 317 nmol/L [≥ 140 ng/mL]) as assessed by the local laboratory during screening (supplementation and retest during screening is acceptable)
* Adequate vitamin B12 (≥ 148 pmol/L [≥ 200 pg/mL]) as assessed by the local laboratory during screening (supplementation and retest during screening is acceptable)
* 18 years of age or older
* Subject or subject's legally acceptable representative has provided informed consent -

Exclusion Criteria:

* Previously diagnosed with intermediate-2 or high risk MDS per IPSS
* Therapy-related or secondary MDS
* History of acute leukemia
* Evidence of bone marrow collagen fibrosis
* Inherited anaemia (eg, haemoglobinopathy, thalassemia, red cell membrane defect, red cell enzyme deficiency), active hemorrhage, red cell aplasia, haemolytic anaemia
* History of malignancies other than curatively treated non-melanoma skin or in situ carcinoma
* History of thrombosis within 6 months prior to randomisation
* Previous bone marrow or stem cell transplantation
* Uncontrolled angina, uncontrolled heart failure, or uncontrolled cardiac arrhythmia as determined by the investigator at screening. Subjects with known myocardial infarction within 6 months prior to randomisation
* Uncontrolled hypertension defined as systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg at screening
* Clinically significant systemic infection or uncontrolled chronic inflammatory disease (ie, rheumatoid arthritis, inflammatory bowel disease) as determined by the investigator at screening
* History of seizure disorder (subject with previous history of seizure disorder will be eligible for the study if he/she had no evidence of seizure activity within 5 years of randomisation and is currently free of antiseizure medication)
* Previous or ongoing use of erythropoiesis-stimulating agent (ESA) therapy, eg, recombinant human erythropoietin (rHuEpo), darbepoetin alfa
* High transfusion demand: receiving a total of ≥ 4 units of RBC transfusion during either of 2 consecutive 8-week periods (ie, days -113 to -57 or days -56 to 0) prior to randomisation
* Received any RBC transfusion within 14 days prior to randomisation
* Received cytotoxic chemotherapy for any oncologic indication or planning to receive cytotoxic chemotherapy during the double-blind treatment period of the study
* Received biologic response modifiers (eg, thalidomide, lenalidomide, arsenic trioxide, azacitidine, decitabine) to treat MDS or planning to receive biologic response modifiers during the double-blind treatment period of the study
* Received myeloablative or craniospinal radiation or planning to receive myeloablative or craniospinal radiation during the double-blind treatment period of the study
* Received granulocyte colony stimulating factor (G-CSF) therapy within 30 days prior to randomization or planning to receive G-CSF therapy during the double-blind treatment period of the study (temporary use of G-CSF for neutropenia with fever and/or infection is acceptable)
* Abnormal renal function (serum creatinine level > 2 times the upper limit of the respective normal range [ULN]) as assessed by the central laboratory at screening
* Abnormal liver function (total bilirubin > 2 times, alanine aminotransferase [ALT] or aspartate aminotransferase [AST] > 3 times ULN) as assessed by the central laboratory at screening. (Subjects with abnormal bilirubin at screening due to documented Gilbert's Disease are eligible if all other criteria are met.)
* Serum endogenous erythropoetin (EPO) level > 500 mU/mL as assessed by the central laboratory at screening
* Known seropositivity for human immunodeficiency virus (HIV) or diagnosis of acquired Immunodeficiency syndrome (AIDS), positive for hepatitis B surface antigen, or seropositive for hepatitis C virus
* Subjects with active ethanol abuse, as judged by the investigator
* Currently enrolled in another investigational device or drug study, or less than 30 days since ending another investigational device or drug study(s), or receiving other investigational agent(s)
* Female subject is not willing to use highly effective contraception during treatment and for at least 1 month after the end of treatment
* Female subject is pregnant or planning to become pregnant within 1 month after the end of treatment
* Subject has known sensitivity to any of the products to be administered during dosing
* Subject has previously been randomised into this study
* Subject will not be available for protocol-required study visits, to the best of the subject and investigator's knowledge
* Subject has any kind of disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or to comply with all required study procedures
* Confirmed history of neutralising antibody activity to rHuEpo or darbepoetin alfa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2011-12-21 (Actual); Primary Completion 2015-02-11 (Actual); Study Completion 2017-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (66):
- Austria (4):
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
- Belgium (11):
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Ghent
  - Research Site, Haine Saint Paul - La Louviere
  - Research Site, Hasselt
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Ottignies
  - Research Site, Roeselare
  - Research Site, Sint-Niklaas
- Czechia (6):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Ostrava-Poruba
  - Research Site, Prague
  - Research Site, Zlín
- France (11):
  - Research Site, Avignon
  - Research Site, Bobigny
  - Research Site, Caen
  - Research Site, Lyon
  - Research Site, Lyon Cédex 3
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Pontoise
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
- Germany (9):
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Göttingen
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, Mannheim
  - Research Site, Regensburg
  - Research Site, Rotenburg (Wümme)
  - Research Site, Ulm
- Greece (4):
  - Research Site, Athens
  - Research Site, Ioannina
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Italy (13):
  - Research Site, Alessandria
  - Research Site, Bologna
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Palermo
  - Research Site, Pavia
  - Research Site, Pesaro
  - Research Site, Pisa
  - Research Site, Reggio Calabria
  - Research Site, Rionero in Vulture PZ
  - Research Site, Roma
  - Research Site, San Giovanni Rotondo FG
  - Research Site, Udine
- Spain (4):
  - Research Site, Zaragoza, Aragon
  - Research Site, Salamanca, Castille and León
  - Research Site, Barcelona, Catalonia
  - Research Site, Valencia, Valencia
- Switzerland (4):
  - Research Site, Basel
  - Research Site, Lucerne
  - Research Site, Muensterlingen
  - Research Site, Zurich

REFERENCES:
- [Background] Platzbecker U, Symeonidis A, Oliva EN, Goede JS, Delforge M, Mayer J, Slama B, Badre S, Gasal E, Mehta B, Franklin J. A phase 3 randomized placebo-controlled trial of darbepoetin alfa in patients with anemia and lower-risk myelodysplastic syndromes. Leukemia. 2017 Sep;31(9):1944-1950. doi: 10.1038/leu.2017.192. Epub 2017 Jun 19. PMID 28626220
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 49 centers in 9 countries. Participants were enrolled from 21 December 2011 to 06 January 2014.
  Results are reported for the double-blind treatment period of the study, with a 07 October 2015 data cut-off; the study is ongoing.
Pre-assignment Details: Eligible participants were randomized in a 2:1 ratio to receive darbepoetin alfa or placebo. Randomization was stratified by International Prognostic Scoring System (IPSS) category (low vs intermediate-1 risk) established at screening.
Groups:
- Placebo: Participants received placebo subcutaneous injection every 3 weeks (Q3W) for 24 weeks.
- Darbepoetin Alfa: Participants received darbepoetin alfa 500 µg Q3W for 24 weeks.
Period: Overall Study
Arm/Group | Placebo | Darbepoetin Alfa
Started | 49 | 98
Received Treatment | 49 | 97
Completed | 39 (Completed treatment in the double-blind treatment period) | 87 (Completed treatment in the double-blind treatment period)
Not Completed | 10 | 11
Not completed — Noncompliance | 1 | 0
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Administrative Decision | 0 | 1
Not completed — Death | 2 | 1
Not completed — Other | 1 | 1
Not completed — Protocol-specified Criteria | 1 | 2
Not completed — Discontinued Without Receiving Treatment | 0 | 1

BASELINE CHARACTERISTICS:
Population: Primary Analysis Set includes all randomized and consented participants who received at least 1 dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Darbepoetin Alfa | Total
Number analyzed (Participants) | 49 | 97 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (9.3) | 72.4 (9.4) | 72.4 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 46 | 66
  Male | 29 | 51 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — French clinical sites, per regulation, did not complete the ethnicity question.
  Participants
    Hispanic or Latino | 1 | 2 | 3
    Not Hispanic or Latino | 45 | 90 | 135
    Unknown or Not Reported | 3 | 5 | 8
Race/Ethnicity, Customized [Number; unit: participants]
  White | 49 | 97 | 146
IPSS Risk Category [Number; unit: participants] — The Myelodysplastic Syndrome (MDS) IPSS score assesses the severity of MDS based on 3 prognostic factors each assigned a score: the percentage of bone marrow blasts, chromosome changes in the marrow cells (karyotype) and the presence of one or more low blood cell counts (cytopenias). The IPSS score is the sum of the bone marrow blast + karyotype + cytopenia score and ranges from 0 (low risk) to 3.5 (high risk). Prognosis is categorized as Low risk (score = 0), Intermediate-1 (score 0.5 to 1.0), Intermediate-2 (score 1.5 to 2.0) or High risk (score ≥ 2.5).
  participants
    Low | 25 | 49 | 74
    Intermediate-1 | 24 | 48 | 72
World Health Organization (WHO) Classification of MDS [Number; unit: participants] — The World Health Organization (WHO) classification recognizes eight subtypes of MDS that are distinguished by the percentage of myeloblasts, presence or absence of ringed sideroblasts (i.e., erythroid precursors with iron deposits surrounding the nucleus), presence of a monocytosis or a deletion 5q.
  participants
    Refractory anemia (RA) | 13 | 9 | 22
    RA with ringed sideroblasts (RARS) | 4 | 17 | 21
    Refractory cytopenia multilineage dysplasia (RCMD) | 19 | 45 | 64
    MDS, unclassified (MDS-U) | 1 | 1 | 2
    MDS associated with isolated del(5q) | 2 | 11 | 13
    Refractory anemia with excess blasts-1 (RAEB-1) | 10 | 13 | 23
    Refractory anemia with excess blasts-2 (RAEB-2) | 0 | 0 | 0
    Unknown | 0 | 1 | 1
Time since MDS Diagnosis [Mean (Standard Deviation); unit: months] — Data available for 43 and 88 participants in each treatment group respectively
  months | 11.7 (17.6) | 12.4 (16.7) | 12.2 (16.9)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] — Data available for 35 and 75 participants in each treatment group respectively
  g/dL | 9.10 (0.87) | 9.23 (0.70) | 9.19 (0.76)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Red Blood Cell (RBC) Transfusion During the Double-blind Treatment Period
Time Frame: Week 5 to Week 25
Population: Transfusion Primary Analysis Set which includes all randomized and consented participants who received at least 1 dose of study drug and who had an end of treatment period (EOTP) visit ≥ day 29 (ie, start of week 5).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 49 | 97
percentage of participants | 59.2 | 36.1
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; The primary hypothesis to be tested was that the percentage of participants with at least 1 RBC transfusion from week 5 to the EOTP was lower in the darbepoetin alfa group than in the placebo group. This hypothesis was confirmed if the incidence of RBC transfusion in the darbepoetin alfa group was lower and had a p-value < 0.05 from a 2-sided Chi-square test; Test type: Superiority or Other; p = 0.008, Chi-squared

2. Secondary Outcome: Percentage of Participants Who Achieved an Erythroid Response Based on International Working Group (IWG) 2006 Criteria in the Double-blind Treatment Period
Description: International Working Group 2006 erythroid response was defined as achieving an initial ≥ 1.5 g/dL increase in hemoglobin from baseline and sustaining an average rise of ≥ 1.5 g/dL in a rolling 56-consecutive day period in the absence of RBC transfusion.
  Participants with no hemoglobin collected to the minimum time required to observe an IWG erythroid response (Week 13) were considered non-responders.
Time Frame: Up to 24 weeks
Population: Primary analysis set participants with a central laboratory baseline hemoglobin value
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 35 | 75
percentage of participants | 0.0 [0.00 to 10.00] | 14.7 [7.56 to 24.73]
Statistical Analysis 1: Comparison: Placebo vs Darbepoetin Alfa; If the primary hypothesis was confirmed, the secondary hypothesis to be tested was that the percentage of participants achieving an IWG erythroid response during the 24-week double-blind treatment period was greater in the darbepoetin alfa group than in the placebo group. This hypothesis was confirmed if erythroid response was higher in the darbepoetin alfa group and the p-value was < 0.05 from a 2-sided Cochran-Mantel-Haenszel test using the IPSS as a stratification factor; Test type: Superiority or Other; p = 0.017, Cochran-Mantel-Haenszel; The overall 2-sided CMH test with IPSS score as stratification factor

3. Secondary Outcome: Number of Participants With Adverse Events
Description: The severity of each adverse event was graded using the the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 grading scale, where grade 1 = mild, grade 2 = moderate, grade 3 = severe, grade 4 = life-threatening and grade 5 = death.
  Prespecified adverse events of interest for darbepoetin alfa, based on clinical data in anemic patients with cancer, included the following categories: hypersensitivity, cardiac failure, hypertension, malignancies, embolic and thrombolic events, venous thromboembolic events (VTEs), central nervous system vascular disorders, and ischemic heart disease.
Time Frame: From first dose of study drug until the end of the double-blind treatment period; 24 weeks.
Population: Safety Analysis Set, including all participants who received at least 1 dose of study drug. One participant in the placebo arm inadvertently received a dose of darbepoetin alfa and is counted in the darbepoetin alfa group for safety analyses.
Measure: Number; unit: participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 48 | 98
participants
  Any adverse event (AE) | 37 | 80
  AE Grade ≥ 2 | 23 | 42
  AE Grade ≥ 3 | 13 | 15
  AE Grade ≥ 4 | 6 | 5
  Serious adverse events (SAE) | 8 | 11
  AE leading to discontinuation of study drug | 2 | 3
  Fatal adverse events | 2 | 1
  Adverse events of special interest | 13 | 16
  Treatment-related adverse events (TRAE) | 4 | 5
  Treatment-related serious adverse events | 0 | 1
  TRAE leading to discontinuation of study drug | 0 | 1
  Treatment-related fatal adverse events | 0 | 0

4. Secondary Outcome: Number of Participants With Disease Progression to Acute Myeloid Leukemia (AML)
Description: Transformation to AML was assessed according to WHO guidelines in the absence of IP and any haematopoietic growth factors (2 weeks off dosing). Bone marrow and/or cytogenetic report confirmation of AML was required (marrow or peripheral blast cells ≥ 20%, presence of pathognomic AML cytogenetic change, or evidence of marrow blast criteria for erythroleukemia). A pathology report confirming other leukemias such as chloroma (granulocytic sarcoma, myeloid sarcoma) or leukemia cutis also constituted transformation to AML.
Time Frame: 24 weeks
Population: Safety analysis set with available data
Measure: Number; unit: participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 46 | 95
participants | 1 | 2

5. Secondary Outcome: Number of Participants With Malignancies Other Than AML, Basal Cell Carcinoma, or Squamous Cell Carcinoma of the Skin
Time Frame: Up to 24 weeks
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 48 | 98
participants | 0 | 1

6. Secondary Outcome: Number of Participants Who Developed Neutralizing Antibodies to Darbepoetin Alfa
Description: Two validated assays were used to detect the presence of anti-darbepoetin alfa antibodies.
  Samples were first tested in an immunoassay to detect antibodies capable of binding to darbepoetin alfa. Samples confirmed to be positive for binding antibodies were subsequently tested in a cell-based assay to determine neutralizing activity against darbepoetin alfa. If a sample was positive for binding antibodies and demonstrated neutralizing activity at the same time point, the sample was defined as positive for neutralizing antibodies.
  The number of participants who developed antibodies to darbepoetin alfa is defined as participants who were neutralizing antibody positive post-baseline with a negative or no result at baseline.
Time Frame: Baseline and end of double-blind treatment period (24 weeks)
Population: Safety analysis set participants with post-baseline antibody results
Measure: Number; unit: participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 43 | 91
participants | 0 | 0

7. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F)
Description: The FACIT-Fatigue scale was a 13-item self-administered questionnaire that assesses both the physical and functional consequences of fatigue. Each question is answered on a 5-point scale, where 0 means "not at all," and 4 means "very much." The FACIT-Fatigue scale score ranges from 0 to 52, with higher scores denoting lower levels of fatigue.
  A positive change from baseline score indicates an improvement. End of treatment period (EOTP) analysis includes last available values.
Time Frame: Baseline, and weeks 13 and 25
Population: FACIT-Fatigue Analysis Set, includes all participants in the primary analysis set who completed or partially completed both the baseline and at least 1 subsequent FACIT-F questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 42 | 90
units on a scale
  Baseline (N = 42, 90) | 32.9 (11.4) | 33.1 (11.4)
  Change from Baseline to Week 13 (n = 41, 85) | -0.9 (9.0) | 2.7 (7.2)
  Change from Baseline to Week 25 (n = 39, 85) | 0.6 (5.5) | 1.2 (8.9)
  Change from Baseline to EOTP (n = 42, 90) | -0.5 (7.1) | 1.1 (8.8)

8. Secondary Outcome: Change From Baseline in EuroQol-5D (EQ-5D) Visual Analog Scale (VAS)
Description: The EQ-5D visual analog scale (VAS) is a global evaluation of overall health state with scores ranging from 0 (worse health state a participant can imagine) to 100 (best health state a participant can imagine).
  End of treatment period (EOTP) analysis includes last available values.
Time Frame: Baseline, and weeks 13 and 25
Population: The EQ-5D visual analog analysis set includes all participants in the primary analysis set who completed both the baseline and at least 1 subsequent visual analog scale.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 42 | 90
units on a scale
  Baseline (N = 42, 90) | 64.4 (17.9) | 64.8 (17.2)
  Change from Baseline to Week 13 (n = 41, 83) | -1.9 (15.5) | 2.9 (13.0)
  Change from Baseline to Week 25 (n = 39, 81) | 2.1 (15.3) | 2.4 (13.5)
  Change from Baseline to EOTP (n = 42, 89) | 0.8 (15.7) | 2.1 (13.1)

9. Secondary Outcome: Percentage of Participants With a Clinically Meaningful Improvement in Fatigue
Description: The FACIT-Fatigue scale was a 13-item self-administered questionnaire that assesses both the physical and functional consequences of fatigue. Each question is answered on a 5-point scale, where 0 means "not at all," and 4 means "very much." The FACIT-Fatigue scale score ranges from 0 to 52, with higher scores denoting lower levels of fatigue.
  Clinically meaningful improvement in fatigue is defined as an increase of ≥ 3 points in the FACIT-Fatigue subscale score, from baseline to EOTP.
Time Frame: Baseline to week 24
Population: FACIT-fatigue analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Darbepoetin Alfa
Number analyzed (Participants) | 42 | 90
percentage of participants | 31.0 [17.62 to 47.09] | 35.6 [25.74 to 46.35]

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 24 weeks for participants who continued into the active treatment period or until 30 days after last dose (maximum of 28 weeks) for participants who did not continue.
Description: One participant randomized to the Placebo arm inadvertently received one 200 µg dose of darbepoetin alfa and is reported in the Darbepoetin alfa group for adverse events.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Darbepoetin Alfa
Serious Adverse Events (participants affected / at risk) | 8/48 | 11/98
Other Adverse Events (participants affected / at risk) | 25/48 | 56/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=48) | Darbepoetin Alfa (N=98)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Proctitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Abscess of salivary gland (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=48) | Darbepoetin Alfa (N=98)
Asthenia (General disorders) | 5 | 12
Fatigue (General disorders) | 4 | 17
Oedema peripheral (General disorders) | 4 | 3
Pyrexia (General disorders) | 1 | 9
Nasopharyngitis (Infections and infestations) | 3 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 5
Dizziness (Nervous system disorders) | 3 | 5
Headache (Nervous system disorders) | 1 | 7
Insomnia (Psychiatric disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.